CLINICAL TRIAL: NCT02718755
Title: Phase II Study of Fludarabine, Cytarabine (ARA-C) and Erwinase IV in Patients With Relapsed or Refractory Hematologic Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Problem with drug supply
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0807; NCI-2016-00691 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Hematologic Malignancy
Keywords: Hematologic malignancy; Relapsed and refractory hematologic malignancies; Acute myeloid leukemia; AML; Acute lymphoblastic leukemia; ALL; Burkitt's leukemia/lymphoma; Prolymphocytic leukemia; Biphenotypic acute leukemia; Blast-phase of chronic myeloid leukemia; CML; B-cell lymphoma; Richter's transformation of chronic lymphocytic leukemia; CLL; Fludarabine; Fludarabine phosphate; Fludara; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma; Leukemia, Prolymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, B-Cell | interventions — fludarabine; fludarabine phosphate; Cytarabine; Asparaginase; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cytarabine + Erwinase (Experimental): Induction Phase: Participants receive 1-2 cycles during the Induction phase.
  Participants receive 1-2 cycles during the Induction phase.
  Participants receive Fludarabine by vein on Days 1-5 and Cytarabine by vein.
  Participants receive Erwinase by vein or as an injection into the muscle on Days 1-7.
  Consolidation Phase: Participants receive up to 3 cycles during the Consolidation phase.
  Participants receive Fludarabine by vein on Days 1-4 and Cytarabine by vein.
  On Day 1 and then every other day for 15 days (3, 5, 7 and so on), participant receives Erwinase by vein or as an injection into the muscle.
  Interventions: Drug: Fludarabine; Drug: Cytarabine; Drug: Erwinase

INTERVENTIONS:
Drug: Fludarabine — Induction Phase:
  30 mg/m2 by vein over 15-30 minutes on Days 1 - 5 of a 28 day cycle.
  Consolidation Phase:
  30 mg/m2 by vein over 15-30 minutes on Days 1 - 4 of a 28 day cycle.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cytarabine — Induction Phase:
  2 grams/m2 by vein over approximately 2 hours on Days 1 - 5 of a 28 day cycle.
  Consolidation Phase:
  2 grams/m2 by vein over approximately 2 hours on Days 1 - 4 of a 28 day cycle.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Erwinase — Induction Phase:
  25,000 Units/m2 by vein (or intramuscularly) over 90-120 minutes on Days 1 - 7 of a 28 day cycle.
  Consolidation Phase:
  25,000 Units/m2 by vein (or intramuscularly) over 90-120 minutes every other day on Days 1, 3, 5, 7, 9, 11, 13, 15 of a 28 day cycle.
  Other Names: L-asparaginase; Erwinia L-Asparaginase; Erwinia Chrysanthemi L-asparaginase

SUMMARY:
The goal of this clinical research study is to learn if fludarabine, cytarabine (ARA-C), and erwinase (also known as asparaginase [erwinia]) in combination can help to control relapsed or refractory hematologic malignancies. The safety of these drugs will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

Each cycle is 28 days.

If participant is found to be eligible to take part in this study, they will receive treatment in 2 phases: Induction and Consolidation.

All participants will receive the same dose level of fludarabine, cytarabine, and erwinase. If the doctor thinks it is needed, the study drug doses may be reduced.

Induction Phase:

Participant will receive 1-2 cycles during the Induction phase.

On Days 1-5, participant will receive fludarabine by vein over about 30 minutes and cytarabine by vein over about 2 hours.

On Days 1-7, participant will receive erwinase by vein over about 2 hours or as an injection into the muscle.

If the disease does not respond during Cycle 1, participant may be allowed to receive an additional Induction cycle. If the disease does respond to Induction, participant can move to the Consolidation phase.

Consolidation Phase:

Participant will receive up to 3 cycles during the Consolidation phase.

On Days 1-4, participant will receive fludarabine by vein over about 30 minutes and cytarabine by vein over about 2 hours. If the doctor thinks it is needed, this may be reduced to Days 1-3.

On Day 1 and then every other day for 15 days (3, 5, 7 and so on), participant will receive erwinase by vein over about 2 hours or as an injection into the muscle.

Study Visits:

On Day 1 (± 3 days) of every cycle, participant will have a physical exam.

Induction Cycle(s):

Every week, blood (about 2-3 teaspoons) will be drawn for routine tests.

On Days 1, 8, 9, and 12 of Cycle 1:

* Blood (about 1-2 teaspoons) will be drawn for routine, biomarker, and pharmacodynamic (PD) testing. Biomarkers are found in the blood/tissue and may be related to how the leukemia reacts to the study drug. PD testing measures how the level of study drug in participant's body may affect the disease.
* On Days 9 and 12 only, blood (about 1-2 teaspoons) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.

On Day 7 of Cycle 1, blood (about 1-2 teaspoons each time) will be drawn for PK testing before the dose and then 8 more times over the next 24 hours after the dose. Some of these blood samples will also be used for antibody testing. Antibodies are created by the immune system and may attack foreign cells or substances, such as the study drug.

On Day 21 of Cycle 1, participant will have a bone marrow aspiration/biopsy for biomarker and PD testing and to check the status of the disease. If the doctor thinks it is needed, participant may have additional bone marrow aspirations/biopsies while on study.

If participant has a second Induction Cycle and the doctor thinks it is needed, they will have a bone marrow aspirate/biopsy at the end of the second Induction Cycle for biomarker and PD testing and to check the status of the disease.

Consolidation Cycles:

Every 1-2 weeks, blood (about 2-3 teaspoons) will be drawn for routine tests.

On Day 1 of Cycle 1, blood (about 1-2 teaspoons) will be drawn for PK testing before the dose and then 8 more times over the next 24 hours after the dose. Some of this blood sample will also be used for antibody testing.

If participant did not have 2 induction cycles, at the end of Cycle 1 of Consolidation, if the doctor thinks it is needed, they will have a bone marrow aspirate/biopsy for biomarker and PD testing and to check the status of the disease.

Length of Treatment:

Participant may continue taking the study drugs for up to 3 cycles of Consolidation after Induction. Participant will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation in the study will be over after the follow-up visits.

Follow-Up Visits:

Every 4-8 weeks after participant's last dose of study drugs, blood (about 2-3 teaspoons) will be drawn for routine tests.

Every 6-12 months after the last dose of study drugs, the study staff will check on how participant is doing. This will either be done by phone or during a regularly scheduled clinic visit. If participant is contacted by phone, the phone call should last about 10 minutes.

This follow-up will last until participant withdraws from the study or the study ends.

Long-Term Follow-Up:

After patient's participation in this study is over, they will be given the option to enroll in a long-term follow-up study (DR09-0223). Participant's doctor will explain this to them in more detail, and they will be required to sign a separate consent form.

This is an investigational study. Fludarabine and cytarabine are FDA approved and commercially available for the treatment of leukemia. Erwinase is FDA approved and commercially available for use in acute lymphoblastic leukemia. Its use in this study is investigational. The combination of these drugs is investigational. The study doctor can explain how the study drugs are designed to work.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of relapsed or refractory hematologic malignancy including, but not limited to Acute myeloid leukemia (AML), Acute lymphoblastic leukemia (ALL), Burkitt's leukemia/lymphoma, Prolymphocytic leukemia, Biphenotypic acute leukemia, Blast-phase of chronic myeloid leukemia (CML), B-cell lymphoma, or Richter's transformation of chronic lymphocytic leukemia (CLL)
2. Age </= 60 years.
3. Adequate organ function as defined below: liver function (bilirubin < 2mg/dL, AST and/or ALT <2.5 x upper limits of normal (ULN)), kidney function (creatinine < 1.5 x ULN ), known cardiac ejection fraction of > or = 45% within the past 3 months

Eastern Cooperative Oncology Group (ECOG) performance status of </= 2.

5) A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.

6) Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.

7) Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patient with documented hypersensitivity to any of the components of the chemotherapy program.
4. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.
5. Patients with history of clinically significant venous thromboembolism.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Overall Response of Fludarabine, Cytarabine, and Erwinase in Refractory/Relapsed Hematologic Malignancies | 56 days
  Response assessed according to the Revised Recommendations of the International Working Group Response Criteria in Acute Myeloid Leukemia.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) of Fludarabine, Cytarabine, and Erwinase in Refractory/Relapsed Hematologic Malignancies | 21 days
  DFS calculated from date of remission until the date of first objective documentation of disease-relapse or death.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org